CLINICAL TRIAL: NCT05483595
Title: An Examination of Blinding for Chinese Herbal Oral Liquid and Matched Placebo: A Randomized Double-blind Clinical Trial
Brief Title: An Examination of Blinding for Chinese Herbal Oral Liquid and Matched Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BE2022-187
Record Dates: First submitted 2022-07-31; First posted 2022-08-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-09

CONDITIONS: Placebo Evaluate
Keywords: Traditional Chinese medicine; blinding; physical consistency; evaluation method
MeSH Terms: interventions — Prescriptions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZFXN group (Other): Subjects actually testing ZFXN
  Interventions: Drug: Chinese herbal medicine FYTF-919
- Placebo group (Other): Subjects actually testing placebo
  Interventions: Drug: Chinese herbal medicine FYTF-919

INTERVENTIONS:
Drug: Chinese herbal medicine FYTF-919 — Oral liquid 10ml
  Other Names: Zhong Feng Xing Nao (ZFXN) prescription

SUMMARY:
TCM is an essential context of the ICH management in Chinese culture. Given the potential benefits of Chinese herbal medicine Zhongfengxingnao formula (ZFXN) in reducing haematoma and bleeding after acute intracerebral hemorrhage (ICH) from fundamental research and small clinical studies, more reliable evidence is required to guide ICH treatment using TCM. This study is designed to evaluate the blinding and physical consistency between the investigational drug and placebo in RCT, taking the trial named Chinese herbal medicine in patients with acute intracerebral hemorrhage (CHAIN) as an example. Therefore the blinding of placebo as well as and physical consistency with investigated TCM in CHAIN trial will be determined. In addition, an assessment method for blinding and physical consistency could be developed for subsequent placebo evaluations.

DETAILED DESCRIPTION:
A total of 48 subjects will be divided into two parts for manual scoring, which includes not only the proportion of the discrimination to ZFXN, which is the primary outcome in this study, but also the physical (odor, taste) consistency of the two drugs. The primary outcome was the percentage of ZFXN response. The secondary outcomes included artificial sensory score and intelligent sensory attributes of testing drug.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old;
* 2. No visual, olfactory, taste, cognitive impairment;
* 3. Provide written informed consent by patient (or approved surrogate);

Exclusion Criteria:

* 1. Evaluation personnel involved in the clinical trial about ZFXN;
* 2. Subjects with severe history of heart, liver, kidney, digestive tract, nervous system, respiratory system, mental disorders or metabolic disorders;
* 3. Subject with history of food, drug allergies, or other allergic diseases (asthma, urticaria, eczematous dermatitis, etc.) or is known to be allergic toZFXN;
* 4. Known definite contraindication to the Chinese herbal medicine;
* 5. Women who are known to be pregnant or lactating;
* 6. Subjects not fit to participate in this study judged by responsible treating clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The percentage of ZFXN response | Within 10 minutes after the first test.
  The incidence of judging testing drug as ZFXN

SECONDARY OUTCOMES:
The artificial sensory score of testing drug | Within 10 minutes after the second test.
  Compare the consistency or difference of artificial sensory (odor, taste) score between two drugs. The value range from 0 to 10: higher scores mean a better consistency.
The intelligent sensory attributes of testing drug | Immediately after testing by electronic nose an electronic tongue.
  Compare the consistency or difference of artificial sensory (odor, taste) score between two drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Guangdong Province Hospital of Chinese Medicine, Guangzhou, Guangdong, China